CLINICAL TRIAL: NCT02137941
Title: Stress Management Programs in Fire-fighters of Paris: a Randomized Controlled Trial
Brief Title: Stress Management Programs in Fire-fighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Defence Health Service (Other Government)
Responsible Party: Principal Investigator, Frédéric Dutheil, Dr, University Hospital, Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: n° EudraCT 2010-A00212-37
Record Dates: First submitted 2014-05-02; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Stress; Anxiety
Keywords: Stress; occupations; biomarkers; firefighters
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- techniques to optimize potential (TOP) (Active Comparator)
  Interventions: Behavioral: techniques to optimize potential (TOP)
- heart coherence (HC) (Active Comparator)
  Interventions: Behavioral: heart coherence (HC)
- controls (Placebo Comparator)

INTERVENTIONS:
Behavioral: techniques to optimize potential (TOP) — The TOP consists of learning easy techniques in mental skills to improve cognitive-based problem-solving using respiration, relaxation, and visualization.
  Arms: techniques to optimize potential (TOP)
Behavioral: heart coherence (HC) — The heart coherence (HC) is based on the fact that the heart rhythm becomes more erratic with negative emotions such as anger and anxiety, and more ordered/coherent with sustained positive emotions such as appreciation, love, or compassion, leading to optimal performance and well-being. The HC program uses feedback from a simple pulse sensor to reflect changes of the emotional/psychological state, and to learn how to reduce stress and stabilize emotions.
  Arms: heart coherence (HC)

SUMMARY:
Chronic stress at work is a public health problem increasing morbidity and mortality, especially in men. Among the men military populations, the firefighters of Paris (FFPs) are particularly exposed. To deal with this stress and to improve stress management is challenging. Psychological fitness is required to regulate emotions which improve effectiveness under stress and enhance recovery from stressful events. The heart coherence (HC) program uses feedback from a simple pulse sensor to reflect changes of the emotional/psychological state, and to learn how to reduce stress and stabilize emotions. Another kind of psychological fitness focuses on cognitive training to regulate emotions, with the use of techniques to optimize potential (TOP). The TOP consists of learning easy techniques in mental skills to improve cognitive-based problem-solving using respiration, relaxation, and visualization. Although never published in a peer-review journal, the procedure of TOP training is structured and standardized for individuals and groups, and is widely practiced in air traffic controllers, with apparently good effects.

Moreover, any event can be emotionally ambiguous, providing both negative and positive outcomes. The interpretation of such ambiguity is linked with an individual's emotional state, such as anxiety or mood. Individuals with a high level of trait anxiety are likely to interpret an event negatively.

However, no studies have compared the effect of HC or TOP in the perceived stress of FFPs. Nor have long-term effects of these stress management programs (SMP) been investigated. Furthermore, the influence of trait anxiety on stress levels in FFPs needs to be clarified. Finally, no trials have assessed levels of biomarkers stress following these SMP.

From these observations, we hypothesized that 1) young recruits aiming to become FFPs will be particularly exposed to stress, 2) SMP will be effective in reducing perceived stress, 3) SMP will mainly benefit FFPs who have high anxiety, and 4) the effects of SMP will lower levels of biomarkers of stress.

The aim of this randomized control trial is to evaluate the effectiveness of stress management programs on perceived stress (primary outcome variable), and on negative mood, mindfulness, and biomarkers of stress (secondary outcome variables) in FFPs. We also aim to investigate the influence of anxiety on the stress management programs effectiveness long-term.

DETAILED DESCRIPTION:
The army's FFPs unit recruits new FFPs each month who received a twelve-month contract comprising of a six-month induction program (1st month to 6th month) and a six-month active duty period (6th month to 12th month). Within our study, volunteers will be included at the 4th month (baseline measurements after the first four months of training), in order to avoid the high drop-out rate that occurs during the beginning of this period. Included participants will be randomly assigned (computer-generated randomization) to one of the three following groups: TOP, HC, or control, and the stress managements programs will occur during the last two months of induction program (4th month to 6th month). The two stress managements programs will be taught by an experimented psychologist, with daily requirements of short practice tasks. All three groups will receive a pharmaceutical placebo in order to control any placebo effect. The placebo will comprise of starch concealed in a capsule, and was required to be consumed between the 4th month and the 6th month.

The primary outcome will be perceived stress. Secondary outcomes will be changes in mood, mindfulness and biomarkers of stress.

All baseline assessments (4th month) will be repeated three times: at the end of the stress managements programs (6th month), at the end of the six-month active duty period (12th month) and at the 18th month.

Enrolment will set to end when 180 FFPs (60 per group) will be included. We estimated that with 55 participants in each group, the study would have more than 80% power to detect a clinically important difference among the groups in the change of perceived stress, at an alpha level of 5%.

Gaussian distribution of the data wil be tested by the Kolmogorov-Smirnov test. Data will be presented as mean ± standard deviation (SD). Comparisons between groups will be made with Wilcoxon matched-pairs test or ANOVA when appropriate. Relationships between data will be assessed by Pearson correlation, a Principal Components Analysis or a multivariable generalized estimating equations model when appropriate. Significance will be accepted at the p<0.05 level. Statistical procedures will be performed using SPSS Advanced Statistics software (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* male starting the formation to be a firefighter of Paris

Exclusion Criteria:

* female
* endocrine disease
* recent extraprofessional life stress event (such as death of a near relative, divorce)
* previous psychological training
* current illness
* medications used to modulate inflammatory diseases (corticosteroids, anti-inflammatory drugs, immunomodulatory drugs)
* medications with a chronotropic effect taken over the previous six months (such as beta blockers, diltiazem, verapamil, anxiolytics or antidepressants)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Perceived stress at the end of the stress managements programs | All baseline assessments (4th month) will be repeated three times: at the end of the stress managements programs (6th month), at the end of the six-month active duty period (12th month) and at 18th month.
  Perceived stress scale (PSS)

SECONDARY OUTCOMES:
the profile of mood states (POMS) | 4th month (baseline), 6th month, 12th month, and 18th month
the Freiburg Mindfulness Inventory-14 | 4th month (baseline), 6th month, 12th month, and 18th month
the Spielberger State-Trait-Anxiety Inventory (S-STAI) | 4th month (baseline), 6th month, 12th month, and 18th month
heart rate variability | 4th month (baseline), 6th month, 12th month, and 18th month
salivary cortisol | 4th month (baseline), 6th month, 12th month, and 18th month
salivary immunoglobulin A | 4th month (baseline), 6th month, 12th month, and 18th month
urinary catecholamines | 4th month (baseline), 6th month, 12th month, and 18th month

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Fire Brigade, Paris, Paris, France